CLINICAL TRIAL: NCT04357951
Title: D-cycloserine Augmented Treatment: Enhancing Extinction Learning in Youth With Tic Disorders
Brief Title: D-cycloserine Augmented Treatment for Youth With Tic Disorders
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00210948
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Tourette Syndrome
Keywords: habit reversal training; Comprehensive Behavioral Intervention for Tics; d-cycloserine; behavior therapy
MeSH Terms: conditions — Tourette Syndrome | interventions — Cycloserine; Behavior Therapy

STUDY DESIGN:
Intervention Model Description: This trial will evaluate the feasibility and initial efficacy of behavior therapy augmented with d-cycloserine (DCS) compared to behavior therapy augmented with placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, therapists, investigators, and outcome assessors will all be masked to treatment assignment. Only the study coordinator will be aware of random assignment to treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Behavior Therapy + DCS (Experimental): Youth with TD will receive four, 2-hour long sessions of evidence-based behavior therapy delivered in an intensive format. Participants will arrive an hour early for each session to take the d-cycloserine pill prior to starting each session of behavior therapy. Participants, therapists, and outcome assessors will be masked to pill condition.
  Interventions: Drug: d-cycloserine; Behavioral: Behavior Therapy
- Behavior Therapy + Placebo (Active Comparator): Youth with TD will receive four, 2-hour long sessions of evidence-based behavior therapy delivered in an intensive format. Participants will arrive an hour early for each session to take the placebo pill prior to starting each session of behavior therapy. Participants, therapists, and outcome assessors will be masked to pill condition.
  Interventions: Drug: Placebo pill; Behavioral: Behavior Therapy

INTERVENTIONS:
Drug: d-cycloserine — D-cycloserine is an FDA-approved antibiotic medication that has been shown to enhance extinction learning in several studies. It will be paired with 4 sessions of behavior therapy.
  Arms: Behavior Therapy + DCS
Drug: Placebo pill — A pill placebo serves as an active comparator. It will be paired with 4 sessions of behavior therapy.
  Arms: Behavior Therapy + Placebo
Behavioral: Behavior Therapy — All participants will receive 4 sessions of behavior therapy for tics (e.g., habit reversal training, comprehensive behavioral intervention for tics).

SUMMARY:
This pilot study aims evaluate the feasibility and initial efficacy of behavior therapy augmented by d-cycloserine (DCS) compared to behavior therapy augmented by placebo. After an initial assessment to determine eligibility, youth with TD will be randomly assigned to receive four sessions of behavior therapy augmented by either DCS or placebo. D-cycloserine is an FDA-approved antibiotic medication that has been shown to enhance extinction learning in several studies. The investigators' proof-of-concept work has found that a single session of DCS-augmented behavior therapy reduced the severity of tics targeted in treatment on the Hopkins Motor/Vocal Tic Scale (HM/VTS) compared to placebo-augmented behavior therapy. This highlights the exciting potential of combining DCS with behavior therapy to improve reductions in tic severity. However, prior to a large-scale clinical trial, it is essential to determine the feasibility and efficacy of augmenting behavior therapy with DCS over multiple treatment sessions.

DETAILED DESCRIPTION:
Tourette's Disorder and Persistent Tic Disorders (collectively referred to as TD) are characterized by the presence of motor and/or vocal tics. For many youth with TD, the severity of tics results in considerable functional impairment and a poor quality of life. While historically managed with psychotropic medications, behavior therapy has demonstrated efficacy for reducing the severity of tics. However, only 50% of youth with TD exhibit a positive treatment response to behavior therapy, and many treatment responders continue to experience bothersome tics. Thus, there is a need to investigate strategies to improve therapeutic outcomes from behavior therapy for youth with TD.

This pilot study aims evaluate the feasibility and initial efficacy of behavior therapy augmented by d-cycloserine (DCS) compared to behavior therapy augmented by placebo. After an initial assessment to determine eligibility, youth with TD will be randomly assigned to receive four sessions of behavior therapy augmented by either DCS or placebo. D-cycloserine is an FDA-approved antibiotic medication that has been shown to enhance extinction learning in several studies. The investigators' proof-of-concept work has found that a single session of DCS-augmented behavior therapy reduced the severity of tics targeted in treatment on the Hopkins Motor/Vocal Tic Scale (HM/VTS) compared to placebo-augmented behavior therapy. This highlights the exciting potential of combining DCS with behavior therapy to improve reductions in tic severity. However, prior to a large-scale clinical trial, it is essential to determine the feasibility and efficacy of augmenting behavior therapy with DCS over multiple treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

* 8-17 years
* Meet Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria for Tourette's Disorder, Persistent Motor Tic Disorder, or Persistent Vocal Tic Disorder
* Have moderate tic severity or greater as evidenced by a Yale Global Tic Severity Scale (YGTSS) total score greater than 13 (>9 for children with motor or vocal tics only)
* Be fluent in English

Exclusion Criteria:

* Current diagnosis of substance abuse/dependence
* Lifetime diagnosis of autism spectrum disorder, mania or psychosis
* History of a seizure disorder, kidney disease, or liver disease
* Four or more previous sessions of behavior therapy

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-04-15 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change in Hopkins Motor/Vocal Tic Scale (HM/VTS) score | Pre-treatment (baseline) and 1 Week post-treatment
  Participants can nominate up to five motor and five vocal tics participants deem bothersome on the HM/VTS. Each bothersome tic is then rated by a clinician on a 5-point scale ranging from none (0) to severe (4). The individual tic scores are summed (minimum of 0 and maximum of 40) and averaged together to create an average tic severity score. Lower scores represent less tic severity, and higher scores indicate greater tic severity. The primary outcome will be the difference in the average score of the two bothersome tics on the HM/VTS that were targeted in treatment (range: 0-8). Change scores were calculated by subtracting the average of the two bothersome tics on the HM/VTS at post-treatment from the average of the two bothersome tics on the HM/VTS at the pre-treatment assessment. Positive scores indicate improvement/decrease in targeted tic severity, with negative scores indicating increase in targeted tic severity.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph McGuire, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot study intended to demonstrate feasibility and test preliminary efficacy. The investigators do not plan to share individual participant data.